CLINICAL TRIAL: NCT00062959
Title: Preventing Problem Behaviors Among Middle School Students
Brief Title: Preventing Problem Behavior Among Middle School Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: N01HD33207; Z01 HD 02110-07-PR; NO1-HD-3-3207; NICHD-400; Z01HD002110-07 (NIH)
Record Dates: First submitted 2003-06-18; First posted 2003-06-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-05

CONDITIONS: Substance Use Disorders; Health Promotion
Keywords: Adolescence; Parenting; School; Primary Prevention; School-based intervention
MeSH Terms: conditions — Substance-Related Disorders

INTERVENTIONS:
Behavioral: Going Places: School program to prevent problem behavior

SUMMARY:
Problem behaviors such as drug use, violence, and school misconduct increase during adolescence. This study evaluated a program designed to prevent problem behaviors in middle school students; the program includes classroom instruction for students and home instruction for parents.

DETAILED DESCRIPTION:
The prevalence of problem behaviors, such as school misconduct, underachievement, and dropout; tobacco, alcohol, and other drug use; and violence and delinquency, increases dramatically during adolescence. These behaviors place youths at an increased risk for school failure, involvement in the criminal justice system, and chronic substance abuse.

The purpose of this study was to test the efficacy of a comprehensive program of interventions, called Going Places, that includes participatory classroom curriculum, parent education, and enhanced school environment. The primary goal of these components was to help students learn social competence skills that will help them make positive decisions in their lives. The classroom curriculum component was integrated into the participating schools' regular Language Arts curriculum in grades 6 through 8. The curriculum provided instruction in and opportunities to practice interpersonal communication, self-management, problem solving, and conflict management. Brief videotapes with student actors served as trigger films to stimulate student interest, provide models, and motivate prosocial behavior. Parents in the participating schools received instruction via videotape and print materials and participated in student homework exercises. The emphasis was on encouraging parents to remain involved, adopt creative monitoring practices, and foster adolescent autonomy by establishing rules and conditions leading incrementally to greater independence.

Students in the seven Charles County, Maryland, middle schools were randomized either to the Going Places intervention group or to the usual education control group. The intervention was sequentially structured, with curricula implemented in each grade of middle school. Questionnaires were administered to all middle school students at the beginning of the 6th grade (before the intervention) to establish baseline levels of substance use, school misconduct, parent and peer influences, and school climate. Students completed surveys in the spring of grades 6, 7, and 8. A final follow-up survey was completed in the fall of ninth grade. The surveys assessed standard measures of tobacco, alcohol, and illicit drug use, school misconduct, and participation in school activities. The surveys also included items related to psychosocial, parental, and school factors.

ELIGIBILITY:
Inclusion Criteria

* Attends participating middle schools
* Reads at grade level

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2768
Dates: Start 1994-06; Study Completion 2000-06

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Simons-Morton, EdD, MPH, Principal Investigator — Prevention Research Branch, Division of Epidemiology, Statistics and Prevention Research

REFERENCES:
- [Background] Simons-Morton BG, Crump AD. Association of parental involvement and social competence with school adjustment and engagement among sixth graders. J Sch Health. 2003 Mar;73(3):121-6. doi: 10.1111/j.1746-1561.2003.tb03586.x. PMID 12683346
- [Background] Simons-Morton BG. Prospective analysis of peer and parent influences on smoking initiation among early adolescents. Prev Sci. 2002 Dec;3(4):275-83. doi: 10.1023/a:1020876625045. PMID 12465590
- [Background] Simons-Morton B, Haynie DL, Crump AD, Eitel SP, Saylor KE. Peer and parent influences on smoking and drinking among early adolescents. Health Educ Behav. 2001 Feb;28(1):95-107. doi: 10.1177/109019810102800109. PMID 11213145
- [Background] Simons-Morton BG, Crump AD, Haynie DL, Saylor KE. Student-school bonding and adolescent problem behavior. Health Educ Res. 1999 Feb;14(1):99-107. doi: 10.1093/her/14.1.99. PMID 10537951
- [Background] Simons-Morton B, Crump AD, Haynie DL, Saylor KE, Eitel P, Yu K. Psychosocial, school, and parent factors associated with recent smoking among early-adolescent boys and girls. Prev Med. 1999 Feb;28(2):138-48. doi: 10.1006/pmed.1998.0404. PMID 10048105
- [Background] Simons-Morton B, Haynie DL, Crump AD, Saylor KE, Eitel P, Yu K. Expectancies and other psychosocial factors associated with alcohol use among early adolescent boys and girls. Addict Behav. 1999 Mar-Apr;24(2):229-38. doi: 10.1016/s0306-4603(98)00095-1. PMID 10336104
- [Background] Haynie DL, Nansel T, Eitel P, Crump AD, Saylor K, Yu K, Simons-Morton, B. Bullies, victims, and bully-victims: Distinct groups of youth at risk. Journal of Early Adolescence 21(1):95-107, 2001.